CLINICAL TRIAL: NCT07304089
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of VIM0423 in Individuals With Isolated Dystonia (Stride Dystonia)
Brief Title: A Study to Evaluate the Efficacy, Safety, and Tolerability of VIM0423 in Individuals With Isolated Dystonia
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vima Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VIM0423-201
Record Dates: First submitted 2025-12-22; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Dystonia
Keywords: Dystonia; Isolated Dystonia; Primary Dystonia; Cervical Dystonia; Segmental Dystonia; Multi-focal Dystonia; Generalized Dystonia
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Torticollis

STUDY DESIGN:
Intervention Model Description: Parallel cohorts of participants receiving active or placebo drug products
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study sponsor, participants, the CRO, Investigator, and all site personnel (except pharmacists and pharmacy staff) will be blinded to treatment assignments until the database has been locked and restricted from further edits.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Segmental/multifocal Active (Active Comparator): Segmental/Multifocal isolated dystonia (enrolling participants with at least two body parts affected receiving active n~40
  Interventions: Drug: VIM0423
- Segmental/multifocal Placebo (Placebo Comparator): Segmental/Multifocal isolated dystonia (enrolling participants with at least two body parts affected) receiving placebo n~40
  Interventions: Drug: VIM0423 Placebo
- Generalized Active (Active Comparator): Generalized isolated dystonia (enrolling participants with more than two body parts affected) receiving active n~10
  Interventions: Drug: VIM0423
- Generalized Placebo (Placebo Comparator): Generalized isolated dystonia (enrolling participants with more than two body parts affected) receiving placebo n~10
  Interventions: Drug: VIM0423 Placebo

INTERVENTIONS:
Drug: VIM0423 — VIM0423 is a combination drug product containing two active ingredients (VMA-1001 and VMA-1002)
  Arms: Generalized Active; Segmental/multifocal Active
Drug: VIM0423 Placebo — Matching VIM0423 placebo product containing no active ingredient
  Arms: Generalized Placebo; Segmental/multifocal Placebo

SUMMARY:
Stride Dystonia is a randomized, double-blind, placebo-controlled study to evaluate the efficacy, safety, and tolerability of VIM0423 in individuals with isolated dystonia.

The main objectives of this clinical trial are to determine the following:

* Does VIM0423 therapy improve dystonia symptoms compared to placebo?
* Is VIM0423 well tolerated in individuals with isolated dystonia? and
* Do the therapeutic effects of VIM0423 confer improvements on daily function and quality of life?

DETAILED DESCRIPTION:
Isolated dystonia, previously referred to as primary dystonia, is a rare movement disorder subclassified according to parts of the body affected. Approximately 160,000 individuals in the United States are affected. Dystonia is characterized by sustained muscle contractions which cause abnormal movements and/or postures. These can be patterned, twisting, or tremulous.

Botulinum toxins (BoNT) are the only approved drug products in the US for the treatment of dystonia; however, these injections are only approved for individuals with a diagnosis of cervical (neck) dystonia or blepharospasm (eye lid) and act locally to weaken affected muscles. There are no approved treatment options for approximately 50% of individuals with other subtypes of isolated dystonia that affect more than one body part, and there are no approved oral treatments for dystonia.

VIM0423 is being developed as a once-daily oral medication that will address the root cause of dystonia, which is known to be a chemical imbalance in specific brain regions. As such, VIM0423 is intended to treat most people with isolated dystonia, regardless of the number of body parts affected.

Stride Dystonia (Study VIM0423-201) is a Phase 2, multicenter, randomized, double-blind, placebo-controlled study designed to assess the efficacy, safety, and tolerability of VIM0423 in adults with isolated dystonia that affects two or more body regions. Up to 120 individuals will be enrolled in the trial.

Participants will be randomized (1:1) to receive either VIM0423 or matching placebo (up to 6 pills a day, taken before bed each evening) for 16 weeks. The Investigator and Participant will not know what patients are receiving VIM0423 or placebo, but that information will be available if needed.

The total time of participation in the trial is up to 32 weeks and requires 6 in person visits. The study schedule includes Screening and Baseline (up to 14 weeks, 2 visits), Dose Titration, Dose Maintenance, Dose Taper (16 weeks, 3 Visits), and Safety follow-up (2 weeks, 1 Visit).

Assessments of changes in dystonia including video recordings will be made by study personnel. Clinical labs, EKGs, and Adverse events will be monitored throughout the study. Participants will be asked to perform self-assessments of their dystonia and its impact on their activities of daily living.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be male or nonpregnant female between 18 and 65 years of age (inclusive) at Visit 1 (Screening).
* The participant has a clinical diagnosis of isolated dystonia for at least one year prior to Visit 1 (Screening); has two or more body regions affected by dystonia at Visit 1 (Screening); and has been confirmed by Investigator and Enrollment Authorization Committee.
* The participant may be untreated with BoNT; OR if the participant is being treated with BoNT as part of their standard of care for dystonia, they must meet protocol-specified criteria.
* The participants must meet protocol-specified requirements for baseline scores on the BFM and CGI-S.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Burke-Fahn-Marsden (BFM) Dystonia Rating Scale | From baseline to Week 14
  0-150, higher score worse

SECONDARY OUTCOMES:
Change from baseline in Clinical Global Impression of Severity (CGI-S) as assessed by the clinician | From baseline to Week 14
  1-7, higher score worse
Change from baseline in the Toronto Western Spasmodic Torticollis Rating Scale including head tremor (TWSTRS; as applicable) | From baseline to Week 14
  0-85, higher score worse
Clinical Global Impression of Change (CGI-C) | From baseline to Week 14
  1-7, higher score worse
Patient Global Impression of Change (PGI-C) | From baseline to Week 14
  1-7, higher score worse

OTHER OUTCOMES:
Incidence and severity of treatment emergent adverse events (TEAEs) | From baseline to Week 14

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Vima Site #004, Scottsdale, Arizona
  - Vima Site #019, Englewood, Colorado
  - Vima Site #031, Orlando, Florida
  - Vima Site #007, Olney, Maryland
  - Vima Site #035, Boston, Massachusetts
  - Vima Site #002, Farmington Hills, Michigan
  - Vima Site #020, Philadelphia, Pennsylvania
  - Vima Site #025, Dallas, Texas
  - Vima Site #015, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No